CLINICAL TRIAL: NCT02963961
Title: Cognitive Training for the Prevention of Postoperative Delirium: a Pilot Study
Brief Title: Cognitive Training for the Prevention of Postoperative Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Phillip Vlisides, Assistant Professor, Department of Anesthesiology, University of Michigan Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00119087
Record Dates: First submitted 2016-11-01; First posted 2016-11-15 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Delirium
Keywords: Delirium; Cognition; Prehabilitation; Neuroplasticity
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training (Experimental): Patients will engage in a daily preoperative cognitive training battery (BrainHQ, Posit Science) that aims to improve attention, memory, and visuospatial processing.
  Interventions: Behavioral: Preoperative Cognitive Training Battery
- No Training (No Intervention): Patients will not undergo preoperative cognitive training. Patients will receive standard preoperative care.

INTERVENTIONS:
Behavioral: Preoperative Cognitive Training Battery — Patients will engage in a daily preoperative cognitive training battery (BrainHQ, Posit Science) that aims to improve attention, memory, and visuospatial processing.
  Arms: Cognitive Training

SUMMARY:
Postoperative delirium is a significant public health concern, affecting up to 70% of elderly patients presenting for surgery. Furthermore, postoperative delirium is associated with increased mortality, persistent cognitive decline, increased hospital length of stay, and elevated healthcare costs. Unfortunately, there is a lack of evidence-based strategies that consistently and effectively reduce the risk of delirium. In fact, although the American Geriatrics Society has released guidelines for the prevention of postoperative delirium, the evidence supporting many of the proposed preventive measures has been deemed low quality.

Cognitive training exercises have been shown to improve cognitive function and functional status in community-dwelling elderly adults, and benefits may last for several months to years. Specifically, training exercises have led to improved performance in attention, short-term memory, and visuospatial processing; all of which are implicated as clinical features of delirium. Cognitive training has also strengthened connectivity in brain networks implicated in postoperative delirium. Thus, given these specific neurological benefits afforded, preoperative cognitive training may provide protection against the development of postoperative delirium. As such, the aim of this pilot study is to assess the feasibility of implementing a preoperative cognitive training program for surgical patients at high-risk for delirium and other associated complications.

DETAILED DESCRIPTION:
This will be a single-center study conducted at the University of Michigan Health System. Participants will be prospectively enrolled and randomized to the interventional group (cognitive training) or control group (no training). Recruitment will take place at the University of Michigan Domino's Farms preoperative clinic at least seven days prior to scheduled, elective surgery. The recruitment goal will be 30 patients per group (total N=60) in this feasibility study. A computer-generated, stratified randomization schedule will be utilized.

This study will use an adaptive cognitive training battery that specifically targets attention, working memory, and visuospatial processing (BrainHQ, Posit Science Corporation, San Francisco, CA). These tests have been successfully used across diverse patient populations, demonstrating improvements in cognition and functional outcomes to varying degrees. The level of difficulty of each test is automatically adjusted depending on the participant's performance, with test difficulty increasing as user performance improves. Participants will access the training software platform via home internet connection, and our study team will be able to monitor training progress.

Delirium assessments will be performed using the Confusion Assessment Method, 3-minute diagnostic assessment (3D-CAM) or CAM-ICU as appropriate, and they will take place at baseline, in the postanesthesia recovery unit (PACU), and twice daily from postoperative day (POD) 1-3. The assessor performing the CAM interviews will be blinded to the intervention. Our team has completed formal training in CAM methodology through the NIH-funded (K07AG041835) Center of Excellence for Delirium in Aging: Research, Training, and Educational Enhancement (CEDARTREE) at Beth Israel Deaconess Hospital, Boston, MA.

Cognitive function will be briefly assessed throughout the study period using three tests from the NIH Toolbox Cognition Battery - Flanker Inhibitory Control and Attention Test, List Sorting Working Memory Test, and the Pattern Comparison Processing Speed Test. Collectively, these tests assess executive function, attention, working memory, and processing speed, which are cognitive domains affected by delirium as described above. These tests have been validated in adults up to the age of 85, and they will be administered, via calibrated iPad, to participants at baseline, the morning of surgery, and at the conclusion of the POD3 visit. The purpose of this testing will be to assess for sustained, transferred, cognitive gains afforded by training in the intervention group.

Delirium is a grave public health concern, particularly for surgical patients. Cognitive training has shown promise with improving clinical and neurophysiological traits associated with delirium, though this potential efficacy has not been tested in a preventive manner in vulnerable surgical patients. Cognitive prehabilitation, via targeted cognitive training exercises, may serve as feasible strategy for reducing the risk of delirium its and associated morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years of age and older
* Major noncardiac, non-major vascular, non-intracranial surgery
* Daily access to computer and internet use prior to surgery

Exclusion Criteria:

* Pre-existing cognitive impairment (preoperative delirium and/or not having capacity to provide informed consent)
* Severe auditory or visual impairment
* Emergency surgery
* No daily computer and internet access
* Already participating in cognitive training exercises

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Delirious Patients per Group | By afternoon of postoperative day (POD) 3
  Each participant who has experienced at least one episode of delirium by the postoperative day 3 time point, as determined by daily Confusion Assessment Method (CAM) screening, will then be calculated in each group to provide delirium incidence (%).

SECONDARY OUTCOMES:
Cognitive Function - Attention, Focus | Baseline, immediate preoperative setting, and POD 3
  The Flanker Inhibitory Control and Attention Test from the NIH Toolbox Cognition Battery will be used to assess attention and focus in each study group. Uncorrected standard score (n, 0-10, 0 = no correct answers, 10 = all items answered correctly and with median reaction time 500 milliseconds or faster on each trial) will be reported within individuals to assess for cognitive function change throughout the study period.
Cognitive Function - Memory | Baseline, immediate preoperative setting, and POD 3
  The List Sorting Working Memory Test from the NIH Toolbox Cognition Battery will be used to assess working memory in each study group. Uncorrected standard score (n, 0-26, 0=no items correctly recalled and sequenced, 26=all items correctly recalled and sequenced) will be reported within individuals to assess for cognitive function change throughout the study period.
Cognitive Function - Brain Processing Speed | Baseline, immediate preoperative setting, and POD 3
  The Pattern Comparison Processing Speed Test from NIH Toolbox Cognition Battery will be used to assess brain processing speed in each group. Uncorrected standard score (n, 0-130, 0=no items answered correctly , 130=all items answered correctly) will be reported within individuals to assess for cognitive function change throughout the study period. Age-adjusted and fully adjusted scaled scores (n) will also be reported
Hospital Length of Stay | Length of hospital stay (n = number of days through study completion, up to 30 days) will be assessed in each group
Length of ICU Stay | Length of ICU stay (n = number of days through study completion, up to 30 days) will be assessed in each group
Physical Therapy (PT) Sessions | Within the first 7 days after surgery
  Percentage (%) of prescribed PT sessions participants are able to successfully complete during the first week after surgery

OTHER OUTCOMES:
Pain Severity (1) | PACU through POD3
  Visual Analogue Scale (mm, 0-100, 0 = no pain, 100 = worst pain imaginable)
Pain Severity (2) | PACU through POD3
  Behavioral Pain Scale (n, 3-12, 3 = no pain, 12 = maximum pain)
Postoperative Opioid Administration | PACU through POD3
  Opioid consumption, converted to morphine equivalents (mg) per day

CONTACTS AND LOCATIONS:
Overall Officials: Phillip E Vlisides, MD, Principal Investigator — Department of Anesthesiology - University of Michigan Medical School
Locations (1):
- University of Michigan Medical School, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rebok GW, Ball K, Guey LT, Jones RN, Kim HY, King JW, Marsiske M, Morris JN, Tennstedt SL, Unverzagt FW, Willis SL; ACTIVE Study Group. Ten-year effects of the advanced cognitive training for independent and vital elderly cognitive training trial on cognition and everyday functioning in older adults. J Am Geriatr Soc. 2014 Jan;62(1):16-24. doi: 10.1111/jgs.12607. Epub 2014 Jan 13. PMID 24417410
- [Background] Kundu B, Sutterer DW, Emrich SM, Postle BR. Strengthened effective connectivity underlies transfer of working memory training to tests of short-term memory and attention. J Neurosci. 2013 May 15;33(20):8705-15. doi: 10.1523/JNEUROSCI.5565-12.2013. PMID 23678114
- [Background] Zelinski EM, Spina LM, Yaffe K, Ruff R, Kennison RF, Mahncke HW, Smith GE. Improvement in memory with plasticity-based adaptive cognitive training: results of the 3-month follow-up. J Am Geriatr Soc. 2011 Feb;59(2):258-65. doi: 10.1111/j.1532-5415.2010.03277.x. PMID 21314646
- [Background] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Bauer PJ, Carlozzi NE, Slotkin J, Blitz D, Wallner-Allen K, Fox NA, Beaumont JL, Mungas D, Nowinski CJ, Richler J, Deocampo JA, Anderson JE, Manly JJ, Borosh B, Havlik R, Conway K, Edwards E, Freund L, King JW, Moy C, Witt E, Gershon RC. Cognition assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S54-64. doi: 10.1212/WNL.0b013e3182872ded. PMID 23479546